CLINICAL TRIAL: NCT05700877
Title: Screening and Intervention for Subclinical Coronary Artery Disease in Patients With Type 2 Diabetes: THE STENO INTEN-CT STUDY
Brief Title: Screening and Intervention for Subclinical Coronary Artery Disease in Patients With Type 2 Diabetes
Acronym: STENO INTEN-CT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Per Løgstrup Poulsen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Løgstrup Poulsen, Professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-500143-21-01
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
Keywords: CVD screening
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The Steno Inten-CT study is an investigator-initiated pragmatic open-label event-driven randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are masked for screening results if they are randomized to "standard treatment", but all participants will obtain information on which arm they are randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAC-based treatment (Experimental): Patients randomized to CAC-based treatment, will be stratified into low- or high-risk patients (defined by CAC score=0 or ≥ 100), and hence, allocated to two parallel l clinical studies.
  High-risk patients (CAC≥ 100) in the CAC-based treatment group will be included in a study in which they will receive information on CAC-score, mandatory treatment with dapagliflozin and semaglutide (both study drugs), and advise on further multifactorial treatment of blood lipid levels, blood pressure and antithrombotic therapy.
  Low-risk patients (CAC=0) will be included in a study in which they will receive information on CAC-score and advise on how multifactorial treatment may be de-intensified.
  Interventions: Other: CAC-based treatment strategy
- Standard treatment (Other): Patients randomized to standard treatment and their primary physician are not informed about the screening findings. Patients are encouraged to follow contemporary diabetes guidelines at the time of inclusion. This information will be given in a written letter within a week of randomization.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: CAC-based treatment strategy — The intervention is a combination of screening with a heart CT scan and multifactorial intervention based on the screening results. Participants randomized to CAC-based treatment and with screening results showing high risk of CVD, will receive a multifactorial intervention including the combination of two open label investigational medical products: dapagliflozin 10mg/day and semaglutide 0.25 /week or 0.5 /week or 1.0 /week.
  Arms: CAC-based treatment
Other: Standard treatment — Participants randomized to standard treatment are recommended to follow updated guidelines for CVD prevention.
  Arms: Standard treatment

SUMMARY:
The investigators intend to perform a landmark study to answer whether a combined CVD screening and treatment strategy is beneficial for patients with type 2 diabetes (T2DM) without known cardiovascular disease (CVD)

The investigators aim to answer the following main research questions:

Do screening detected high-risk patients benefit of intensified medical treatment?

Is it safe to de-intensify medical treatment among patients with a screening detected low risk of CVD?

Does a CVD screening and treatment program improve patient reported health status?

Cardiovascular risk remains high in patients with T2DM but unevenly distributed. Our current risk stratification strategies are far from optimal leading to both under- and over-treatment of patients. In recent years, noninvasive imaging of subclinical coronary artery disease by cardiac CT has improved considerably. This allows for easily accessible evaluations of coronary atherosclerosis burden and composition - exceptionally strong imaging biomarkers of future cardiovascular disease. An increasing amount of data suggests that cardiac CT may permit better risk stratification in patients with T2DM. At the same time, the pharmaceutical treatment of T2DM has changed with several new and expensive drug classes, each individually documented to reduce the risk for new or recurrent cardiovascular events. Thus, these new drugs may improve outcome in high-risk patients, whereas they may be wasteful and only lead to side effects in low-risk patients.

In the Inten-CT study, the investigators combine these two pivotal developments. The investigators intend to improve risk stratification of patients with T2DM by use of cardiac CT and, based on this knowledge, the investigators wish to investigate if upgraded medical treatment in the high-risk population is beneficial and if de-intensified treatment in the low-risk population is safe. As a secondary aim, the investigators wish to investigate if such a strategy improves patient reported health status. These aims are in agreement with one of the important health indicators from The Danish College of General Practitioners: "We find and treat the patients and let the healthy stay healthy". The investigators intend with this strategy to improve not only cardiovascular outcome among patients with T2DM, but also their quality of life.

The Inten-CT study is an investigator-initiated open-label event-driven randomized controlled trial including patients with T2DM stratified according to screen detected coronary artery calcification. The investigators expect inclusion of 7300 patients in 2 years and a mean follow-up period of 5 years.

DETAILED DESCRIPTION:
HYPOTHESES Intensified multifactorial treatment is superior to standard treatment in patients with CAC score ≥100.

Less intensive multifactorial treatment is non-inferior to standard treatment in patients with CAC =0.

AIMS Primary aim 1: Cardiovascular benefit In patients identified with high cardiovascular risk as indicated by a CAC score ≥100, the investigators aim to compare the effect of intensified multifactorial treatment versus standard treatment.

Primary aim 2: Cardiovascular safety In patients identified with low cardiovascular risk as indicated by a CAC score of zero, the investigators aim to compare the effect of less intensive multifactorial treatment versus standard treatment.

Secondary aim 1: Patient-reported outcomes the investigators aim to compare patient-reported outcomes in the CAC-based treatment group and the control group.

Secondary outcome: Quality adjusted life years (QALY) using data from the EQ-5D questionnaire and Danish preference weights of the normal population

Secondary aims 2: Cost-Effectiveness The investigators aim to compare costs and outcomes between the two groups after study completion.

Secondary aims 3: Treatment The investigators aim to quantify and compare the protocol-driven and symptom-driven diagnostic tests and therapeutic interventions between the intervention groups and control groups during the study period.

The investigators aim to evaluate the adherence and efficacy of the therapeutic interventions in the intervention groups and the control groups during the study period.

Secondary aims 5: Screening The investigators aim to evaluate the association of CAC score and coronary CT angiography derived measures of coronary atherosclerosis burden, respectively, and CVD prognosis in patients with T2DM.

The investigators aim to explore the association between CAC score, coronary CT angiography derived measures of coronary atherosclerosis burden and echocardiography derived measures of systolic/diastolic function. Specifically, the investigators aim to explore the ability of echocardiography to re-classify patients stratified by CAC and coronary CT angiography.

Secondary aims 6: Biomarkers The investigators aim to explore the association between CAC score, biochemical markers of inflammation and atherosclerosis (blood high-sensitivity C-reactive protein, IL-1ß, IL-6, sE-selectin, sICAM-1, sVCAM, osteopontin, osteoprotegrin and urinary proteomic risk classifier CKD273, CAD258, ACSP75, and HF1), and CVD prognosis in patients with T2DM.

METHODS Design The Steno Inten-CT study is an investigator-initiated pragmatic open-label event-driven randomized controlled trial.

First, a cardiac CT scan is performed in all participants. Next, patients are randomized to either continue standard diabetes treatment blinded to CT scan and CAC results or receive CAC-based treatment. Patients randomized to CAC-based treatment, will be stratified into low- or high-risk patients (defined by CAC score <100 or ≥ 100), and hence, allocated to two parallel clinical studies. High-risk patients in the CAC-based treatment group will be included in a study in which they will receive information on CAC-score, mandatory treatment with dapagliflozin and semaglutide (both study drugs), and advise on further multifactorial treatment of blood lipid levels, blood pressure and antithrombotic therapy. Low-risk patients will be included in a study in which they receive advise on a potential downgrade in diabetes treatment (CAC =0).

Patients with CAC score 1-99 will be advised to follow contemporary guidelines in diabetes treatment and will not be included in the primary analyses (Primary aims 1 and 2).

At End of Study (determined by an independent outcome committee), CVD event rates will be compared between patients in the standard treatment group and the CAC-based treatment group, stratified according to their CAC-level (CAC ≥100, and CAC=0)

ELIGIBILITY:
Inclusion Criteria:

* New or former diagnosis of Type 2 diabetes according to WHO.
* Age between 55-69 years (men) and 60-74 years (women).
* Signed declaration of consent

Exclusion Criteria:

* Previous history of CVD (previous myocardial infarction or coronary intervention (percutaneous coronary intervention or by-pass), heart failure, stroke or peripheral artery disease as documented by the patient or the patient medical record).
* Contraindications or allergies to both SGLT2 inhibitors and GLP-1 analogues.
* Signs of critical cardiac disease: >50% stenosis of left main coronary artery (CT angiography) or left ventricular ejection fraction below 30% (echocardiography). If a CT angiography is not available, a CAC>1000 on the non-contrast cardiac CT will be considered equal to critical cardiac disease.
* Expected life duration < 1 year for any reason.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7300 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Rates of a composite cardiovascular endpoint | Event-driven, expected mean follow-up of 5 years
  Cardiovascular death, non-fatal myocardial infarction, hospitalization for heart failure, and non-fatal stroke

SECONDARY OUTCOMES:
Rates of all-cause mortality and individual components of the primary outcome | Event-driven, expected mean follow-up of 5 years
  Individual components of the primary outcome consist of cardiovascular death, non-fatal myocardial infarction, hospitalization for heart failure, and non-fatal stroke
Patient reported outcomes 1 | Change from baseline to End of Study (Event-driven, expected mean follow-up of 5 years)
  EQ5D questionnaire with the outcome of a EQ5D-score
Patient reported outcomes 2 | Change from baseline to End of Study (Event-driven, expected mean follow-up of 5 years)
  PHQ-9 questionnaire with the outcome of a PHQ-9-score
Patient reported outcomes 3 | Change from baseline to End of Study (Event-driven, expected mean follow-up of 5 years)
  GAD-7 questionnaire with the outcome of a GAD-7-score
Cost-effectiveness | Event-driven, expected mean follow-up of 5 years
  Cost per quality adjusted life years (QALY)

OTHER OUTCOMES:
Treatment with prespecified drugs | Event-driven, expected mean follow-up of 5 years
  Treatment with prespecified CVD prophylactic drugs will be recorded through the national health registries. Treatment initiation will be registered.
Cardiovascular risk markers 1 | Event-driven, expected mean follow-up of 5 years
  Lipid levels (total cholesterol, LDL, HDL and triglycerides) collected in LABKA. Reported as mmol/l
Cardiovascular risk markers 2 | Event-driven, expected mean follow-up of 5 years
  Office blood pressure (mmHg) collected in Dansk Voksen Diabetes Databasen.
Cardiovascular risk markers 3 | Event-driven, expected mean follow-up of 5 years
  Body mass index (kg/m2) collected in Dansk Voksen Diabetes Databasen.
Cardiovascular risk markers 4 | Event-driven, expected mean follow-up of 5 years
  Smoking cessation (number and percentage) collected in Dansk Voksen Diabetes Databasen.

CONTACTS AND LOCATIONS:
Overall Officials: Per L Poulsen, Professor, Principal Investigator — Steno Diabetes Center Aarhus, AUH, and Aarhus University; Axel Diederichsen, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked for consent to participate in a research database and a database for future research. The database will be administered by the Steno DK organization. Rules for external researchers to apply for and access data will be laid out towards the end of the study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: TBA
Access Criteria: TBA

REFERENCES:
- [Derived] Funck KL, Borregaard B, Egstrup K, Fredslund EK, Hansen TW, Kallestrup P, Olsen MH, Reventlow S, Rossing P, Sandbaek A, Sondergaard J, Thomsen JL, Vestergaard P, Poulsen PL, Diederichsen A. Study protocol for the investigator-initiated Danish pragmatic randomised STENO INTEN-CT trial: does screening and intervention for subclinical coronary artery disease in type 2 diabetes reduce cardiovascular events? BMJ Open. 2025 Dec 15;15(12):e106018. doi: 10.1136/bmjopen-2025-106018. PMID 41401988

DOCUMENTS (1):
  • Study Protocol (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT05700877/Prot_000.pdf